CLINICAL TRIAL: NCT01737931
Title: An Open-Label Trial to Explore Symptomatic Therapy for Application Site Reaction to SPM962 in Healthy Subject
Brief Title: A Trial to Explore Symptomatic Therapy for Application Site Reaction to SPM962 in Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 243-12-002
Record Dates: First submitted 2012-11-25; First posted 2012-11-30 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: SPM 962; rotigotine; application site reaction
MeSH Terms: interventions — Steroids; Dexamethasone; Histamine Antagonists; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Topical Steroid (Experimental): Topical medication of steroid (Dexamethasone) to the application sites after the patch removal
  Interventions: Drug: Topical steroid (Dexamethasone)
- Topical antihistamine (Experimental): Topical medication of antihistamine(Diphenhydramine) to the application sites after the patch removal
  Interventions: Drug: Topical antihistamine (Diphenhydramine)
- No-treatment (No Intervention): No treatment to the application sites after the patch removal

INTERVENTIONS:
Drug: Topical steroid (Dexamethasone) — for SPM 962: 1 mg/24h patch for 48 hours as Acceleration period, then 2 mg/24h patch to the other site for 24 hours as Dose-escalation period, for steroid: twice daily administration of Dexamethasone (1 mg/g cream) to the application sites after the patch removal
  Arms: Topical Steroid
Drug: Topical antihistamine (Diphenhydramine) — for SPM 962: 1 mg/24h patch for 48 hours as Acceleration period, then 2 mg/24h patch to the other site for 24 hours as Dose-escalation period, for antihistamine: twice daily administration of Diphenhydramine (10 mg/g cream) to the application sites after the patch removal
  Arms: Topical antihistamine

SUMMARY:
To investigate the efficacy of symptomatic therapy with topical steroids and antihistamines for application site reaction (ASR) after administration of SPM 962 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female and aged between 20 and 45 years of age (inclusive)
* Subject is of normal body weight as determined by a body-mass index (BMI) between 18 and 28 kg/m2
* Subject is healthy as determined by EA (medical history, physical examination, skin evaluation, vital signs, ECG, hematology, clinical chemistry, urinalysis)
* Subject is surgically sterile; subject has been postmenopausal for at least 12 consecutive months if female; or subject agrees to remain abstinent or to follow two acceptable methods of birth control from EA to the end of observation period. (fore male and female subjects)

Exclusion Criteria:

* Subject has a history or complication of epilepsy and/or seizures
* Subject has clinically relevant changes in the ECG, such as second- or third-degree AV block, a complete bundle branch block, prolongation of the QRS complex over 120 ms, or of the QTcB (QT interval corrected for HR by Bazett´s formula) over 500 ms at EA
* Subject has a clinically relevant hepatic dysfunction
* Subject has a clinically relevant renal dysfunction
* Subject has a history of significant skin hypersensitivity to adhesives or other transdermal products or recent unresolved contact dermatitis
* Subject has a history or complication of atopic or eczematous dermatitis, psoriasis, and/or an active skin disease or skin tumors
* Subject has more than 1 known or suspected drug hypersensitivity, in particular to any component of the trial medication
* Subject has a history of chronic alcohol or drug abuse within the last 5 years
* Subject is tested positive for HIV-1/2Ab, HBsAg or HCV-Ab
* Subject tests positive for alcohol and/or drugs at EA
* Subject is taking any prohibited concomitant medication
* Subject has a history or complication of narrow angle glaucoma
* Subject has a history or complication of respiratory or cardiovascular disorders (e.g., heart failure, coronary heart disease, hypertension, arrhythmia, tachyarrhythmia, or myocardial infarction)
* Subject has a history or complication of psychic abnormality, psychiatric or neurologic illness, or autonomic neuropathy
* Subject has a history or complication of diabetes mellitus and/or thyroid dysfunction, especially hyperthyroidism or other endocrine disorders
* Subject has a history or complication of malignancy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Kyeonggi-do
  - Seoul National University Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 120 eligible subjects received the IMP treatment at least once, and 3 of them were withdrawn from the trial before topical treatment allocation due to subject request (1 subject) and for lack of efficacy evaluation (2 subjects).
Period: Overall Study
Arm/Group | Topical Steroid | Topical Antihistamine | No-treatment
Started | 38 | 40 | 39
Completed | 38 | 38 | 38
Not Completed | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Steroid | Topical Antihistamine | No-treatment | Total
Number analyzed (Participants) | 38 | 40 | 39 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (4.2) | 26.7 (4.8) | 26.1 (3.7) | 26.5 (4.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 40 | 39 | 117
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 38 | 40 | 39 | 117
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 38 | 40 | 39 | 117

OUTCOME MEASURES:

1. Primary Outcome: Skin Irritation Score of the Application Site
Description: Skin irritation score of the application site 24 hours after 2 mg/24 hour patch removal (dose-escalation period) and difference between Steroid or Antihistamine and No-treatment.
  The scale scoring criteria are 0(-): Negative, 0.5(±): Faint erythema, 1(+): Erythema, 2(++): Erythema + edema, 3(+++): Erythema + edema + papules, serous papule, vesicles, 4(++++): Coalescing vesicles.
Time Frame: 24 hours after 2 mg/24 hr patch removal
Population: Full analysis set (FAS) subjects with a score of ≥ 0.5 (±) at Day 3
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Topical Steroid | Topical Antihistamine | No-treatment
Number analyzed (Participants) | 19 | 19 | 20
Scores on a scale | 0.237 [0.084 to 0.390] | 0.289 [0.136 to 0.422] | 0.250 [0.101 to 0.399]

2. Primary Outcome: Itching of Application Site Evaluated by the Visual Analogue Scale (VAS)
Description: Itching of application site evaluated by the visual analogue scale (VAS) 24 hours after 2 mg/24 hour patch removal (dose-escalation period) and difference between Steroid or Antihistamine and No-treatment.
  The score ranges from 0 (no itching) to 100 (strongest imaginable itching).
Time Frame: 24 hours after 2 mg/24 hr patch removal
Population: FAS
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Topical Steroid | Topical Antihistamine | No-treatment
Number analyzed (Participants) | 37 | 38 | 38
Scores on a scale | 1.6 [0.5 to 2.7] | 0.4 [-0.7 to 1.6] | 0.9 [-0.2 to 2.0]

3. Secondary Outcome: Skin Irritation Score After Patch Removal
Description: Numbers of subjects with each skin irritation score. The scale scoring criteria are 0(-): Negative, 0.5(±): Faint erythema, 1(+): Erythema, 2(++): Erythema + edema, 3(+++): Erythema + edema + papules, serous papule, vesicles, 4(++++): Coalescing vesicles.
Time Frame: Up to 72 hours after patch removal
Population: FAS subjects with a score of ≥ 0.5 (±) at Day 3
Measure: Number; unit: Percentage of participants
Arm/Group | Topical Steroid | Topical Antihistamine | No-treatment
Number analyzed (Participants) | 19 | 18 | 20
Percentage of participants
  - (1 hour after patch removal) | 5.3 | 5.6 | 10.0
  ± (1 hour after patch removal) | 63.2 | 55.6 | 45.0
  + (1 hour after patch removal) | 31.6 | 38.9 | 45.0
  - (24 hours after patch removal) | 57.9 | 52.6 | 60.0
  ± (24 hours after patch removal) | 36.8 | 36.8 | 30.0
  + (24 hours after patch removal) | 5.3 | 10.5 | 10.0
  - (48 hours after patch removal) | 89.5 | 94.7 | 80.0
  ± (48 hours after patch removal) | 10.5 | 5.3 | 20.0
  - (72 hours after patch removal) | 94.4 | 94.7 | 90.0
  ± (72 hours after patch removal) | 5.6 | 5.3 | 10.0

4. Secondary Outcome: Itching of Application Site Evaluated by VAS After Patch Removal
Description: Changes of itching of application site evaluated by VAS after patch removal (acceleration and dose-escalation periods).
  The score ranges from 0 (no itching) to 100 (strongest imaginable itching).
Time Frame: Up to 96 hours after patch removal
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Topical Steroid | Topical Antihistamine | No-treatment
Number analyzed (Participants) | 38 | 39 | 39
Scores on a scale
  3 hours after patch removal | -2.8 (6.9) | -3.0 (9.0) | -2.2 (4.6)
  6 hours after patch removal | -3.3 (7.9) | -3.3 (8.6) | -2.3 (5.0)
  24 hours after patch removal | -3.9 (10.0) | -2.6 (7.0) | -2.6 (4.7)
  48 hours after patch removal | -3.9 (10.5) | -3.6 (9.0) | -2.9 (5.1)
  72 hours after patch removal | -4.1 (10.0) | -3.8 (8.9) | -3.0 (5.1)
  96 hours after patch removal | -4.3 (10.1) | -3.8 (8.9) | -3.0 (5.1)

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- Over-all: In this study, all the subjects were received SPM962 with the same dose and regimen during the acceleration and dose-escalation periods and then they were randomized into one of the three groups after removal of SPM962 to evaluate recovery of skin reaction caused by SPM962 using either steroids, antihistamine or no treatment.
  Since AEs mainly occurred in the acceleration and dose-escalation periods when SPM962 were used, AEs are shown in one group.
Arm/Group | Over-all
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 41/120
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Over-all (N=120)
Application Site Irritation (General disorders) | 3 (3)
Feeling Hot (General disorders) | 3 (3)
Headache (Nervous system disorders) | 6 (6)
Somnolence (Psychiatric disorders) | 6 (6)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No